CLINICAL TRIAL: NCT05118568
Title: Imaging of Lumpectomy Surface With Large Field-of-View Confocal Laser Scanning Microscope 'Histolog Scanner' for Breast Margin Assessment in Comparison With Intraoperative Imaging and Postoperative Histopathological Assessment
Brief Title: Assessment of Lumpectomy Margins With the Histolog Scanner in Comparison With Intraoperative Imaging Techniques
Acronym: Polarhis
Status: Completed | Type: Observational
Sponsor: SamanTree Medical SA (Industry)
Collaborators: St. Vincenz Krankenhaus GmbH, Paderborn (Unknown)
Responsible Party: Sponsor
Other Study IDs: Polarhis
Record Dates: First submitted 2021-11-01; First posted 2021-11-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Confocal Microscopy; Fresh Tissue Imaging; Intraoperative Assessment; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Histolog Scanner — imaging of fresh lumpectomy specimens with the Histolog Scanner, confocal microscopy scanning medical imaging device

SUMMARY:
Study to assess the capability of using the Histolog Scanner, a recent large field-of-view confocal laser scanning medical imaging device for the breast cancer detection in fresh lumpectomy margins.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. For early-stage breast cancers, breast-conserving surgery (BCS) is applied to excise the tumor while saving surrounding healthy tissue as much as possible to avoid radical excisions and achieve better aesthetic and psychological outcomes for the patient. This surgical approach requires postoperative tumor-free margin assessment of the surgical resection in order to carry on with next steps of the patient care treatment (e.g. radiotherapy). Unfortunately, at least 20% of patient undergo more than one procedure to achieve acceptable margin status due to difficulties to identify subclinical and deep-seated tumor during BCS. During the surgery, the surgeon mainly relies on nonspecific visual changes and manual palpation of subtle irregularities to guide cancer excision. While these determinants enable bulk tumor assessment, they do not offer the information to adequately identify tumor infiltrates on lumpectomy margin.

An efficient intraoperative assessment of the margin may solve these issues and confocal imaging has shown some promises by providing real-time imaging of fresh tissue with the resolution sufficient to visualize microscopic tissue features. The Histolog Scanner is a recent confocal microscope designed for clinical use on large surgical specimens.

The main objective of this study is to confirm that the use of the Histolog Scanner by surgeons allows to detect breast cancer on lumpectomy margins and compare the performance of the detection with local standard-of-care intraoperative imaging techniques (ultrasound and radiography) using the final assessment performed in pathology as reference.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient ≥18 years old
* Patient Scheduled for breast conserving surgery of invasive and/ or in situ ductal carcinoma (DCIS).
* Patient able to read, understand and give informed consent

Exclusion Criteria:

* Patient previously treated for ipsilateral breast cancer surgery
* Patient with previous radiotherapy of the breast
* Patient with multicentric breast cancer
* Patients with planed mastectomy, tumor-adapted breast reduction
* Patient with presurgical neo-adjuvant treatment
* Patient is pregnant/lactating
* Participation in any other clinical study that would affect data acquisition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient are selected by breast surgeons during their standard-of-care preoperative consultations
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Accuracy, Sensitivity, Specificity for breast cancer detection | Through study completion, an average of 6 months
  Quantification of the performance achieved by breast surgeons and pathologists for breast cancer detection in Histolog Scanner images of lumpectomy margins

SECONDARY OUTCOMES:
Theoretical impact on re-operation rates | Through study completion, an average of 6 months
  Extrapolation of the re-operation rate reduction based on positive-margin detection achieved with the Histolog Scanner, in comparison with the local intraoperative margin assessment techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Lux, MD, MBA, Principal Investigator — St. Vincenz-Krankenhaus GmbH
Locations (1):
- St. Vincenz-Krankenhaus GmbH, Frauenklinik St. Louise, Paderborn, Germany